CLINICAL TRIAL: NCT04910867
Title: Integrating a Culturally Competent APOL1 Genetic Testing Program Into Living Donor Evaluation
Brief Title: APOL1 Genetic Testing Program for Living Donors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Elisa Gordon, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DK128207 (NIH)
Record Dates: First submitted 2021-05-08; First posted 2021-06-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases; Apolipoprotein L1; Kidney Transplantation
Keywords: Genetics; Implementation research; Healthcare disparities; Ethics; Informed consent; Safety; African continental ancestry group; genetic counseling; Culturally competent care; Electronic health records; Decision support systems, clinical; Decision making; Live kidney donation; Shared decision making; Artificial intelligence; Surveys and questionnaires; Qualitative research; Clinical trial
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A non-randomized, pre-post design. Data will be collected from participants at both sites during a control period, prior to implementing the intervention, and during an intervention period, under the proposed APOL1 genetic testing program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): No intervention will be administered. Usual care will be administered.
- Intervention Arm (Experimental): APOL1 testing program
  Interventions: Behavioral: Components of Genetic Counseling; Diagnostic Test: APOL1 genetic testing; Other: EHR integration

INTERVENTIONS:
Behavioral: Components of Genetic Counseling — The APOL1 testing program is designed to help living donor candidates to reduce their decisional conflict and enhance their informed consent regarding living donation. This intervention component entails: (1) an artificial intelligence-based conversational agent "chatbot" providing foundational information about the relationship between APOL1 and kidney disease and living donor outcomes, and APOL1 testing. The chatbot helps to relieve the workload on clinicians and scale up information giving. (2) The transplant nephrologist counseling component includes discussion about the APOL1 test results and shared decision making about donation, in a culturally competent manner, so as to enhance donor candidates' informed consent for living donation.
  Arms: Intervention Arm
Diagnostic Test: APOL1 genetic testing — APOL1 genetic testing will be performed while live kidney donor candidates are undergoing donor evaluation to identify whether they are at elevated risk of kidney disease post-donation. This risk information is expected to better enable donor candidates to make meaningful informed decisions about donating.
  Arms: Intervention Arm
Other: EHR integration — APOL1 genetic test results will be integrated into the electronic health record to provide clinical decision support to transplant nephrologists in evaluating donor candidates.
  Arms: Intervention Arm

SUMMARY:
Living donor (LD) kidney transplantation is the optimal treatment for patients with end-stage kidney disease (ESKD). However, LDs take on a higher risk of future ESKD themselves. African American (AA) LDs have an even greater, 3.3-fold, risk of ESKD than white LDs post-donation. Because evidence suggests that Apolipoprotein L1 (APOL1) risk variants contribute to this greater risk, transplant nephrologists are increasingly using APOL1 testing to evaluate LD candidates of African ancestry. However, nephrologists do not consistently perform genetic counseling with LD candidates about APOL1 due to a lack of knowledge and skill in counseling about APOL1. Without proper counseling, APOL1 testing will magnify LD candidates' decisional conflict about donating, jeopardizing their informed consent. Given their elevated risk of ESRD post-donation, and AAs' widely-held cultural concerns about genetic testing, it is ethically critical to protect AA LD candidates' safety through APOL1 testing in a culturally competent manner to improve informed decisions about donating.

No transplant programs have integrated APOL1 testing into LD evaluation in a culturally competent manner. Clinical "chatbots," mobile apps that use artificial intelligence to provide genetic information to patients and relieve constraints on clinicians' time, can improve informed treatment decisions and reduce decisional conflict. The chatbot "Gia," created by a medical genetics company, can be adapted to any condition. However, no chatbot on APOL1 is currently available. No counseling training programs are available for nephrologists to counsel AA LDs about APOL1 and donation in a culturally competent manner. Given the shortage of genetic counselors, increasing nephrologists' genetic literacy is critical to integrating genetic testing into practice.

The objective of this study is to culturally adapt and evaluate the effectiveness of an APOL1 testing program for AA LDs at two transplant centers serving large AA LD populations (Chicago, IL, and Washington, DC). The APOL1 testing program will evaluate the effect of the culturally competent testing, chatbot, and counseling on AA LD candidates' decisional conflict about donating, preparedness for decision-making, willingness to donate, and satisfaction with informed consent. The specific aims are to:

1. Adapt Gia and transplant counseling to APOL1 for use in routine clinical practice
2. Evaluate the effectiveness of this intervention on decisional conflict, preparedness, and willingness to donate in a pre-post design
3. Evaluate the implementation of this intervention into clinical practice by using the RE-AIM framework to longitudinally evaluate nephrologist counseling practices and LDs' satisfaction with informed consent.

The impact of this study will be the creation of a model for APOL1 testing of AA LDs, which can then be implemented nationally via implementation science approaches. APOL1 will serve as a model for integrating culturally competent genetic testing into transplant and other practices to improve patient informed consent.

DETAILED DESCRIPTION:
This project, "Integrating a culturally competent APOL1 genetic testing program into living donor evaluation," will integrate APOL1 testing into the evaluation of living kidney donor candidates of African ancestry. The study aims to reduce decisional conflict, improve preparedness for decision making, and increase satisfaction with informed consent for living donation for donor candidates at elevated risk of post-donation kidney failure. The APOL1 testing program will entail adapting established artificial intelligence conversational agents or "chatbots" to provide APOL1-specific information in preparation for donor candidates to undergo APOL1 testing, and adapting established genetic counseling discussions for transplant nephrologists to counsel donor candidates about APOL1 test results and engage in shared decision making to improve donor candidates' informed consent for living donation. APOL1 test results will be integrated into the electronic health record to provide clinical decision support to transplant nephrologists. The study will involve community engagement to ensure that testing and counseling is delivered in a culturally competent manner.

Using a hybrid effectiveness-implementation design, this study will simultaneously evaluate the effectiveness and implementation of the APOL1 testing program to more efficiently translate evidence into practice, as service delivery system factors for adoption and scale up are considered while effectiveness is tested. The study will be conducted at two geographically distinct transplant programs: Northwestern University in Chicago, IL, and Georgetown University in Washington, DC.

Participants include live kidney donor candidates of African ancestry undergoing donor evaluation. The investigators will recruit potential participants consecutively; with participants recruited in year 1 serving as the control group, and participants recruited in years 2-5 serving as the intervention group. Participants will be eligible for participation if they respond positively to one of three questions assessing African ancestry. Participants in the intervention group will use the chatbot for 5-7 minutes. Immediately thereafter, research staff will ask for participants' informed consent to undergo APOL1 genetic testing; those who agree will provide a saliva sample for testing. APOL1 test results will be integrated into the respective transplant program's electronic health records. Thereafter, transplant nephrologists will engage in a counseling discussion with donor candidates about APOL1 and living donation.

Distributional assumptions will be assessed to evaluate appropriateness of model specifications. For primary analyses, the mixed model framework will allow for incorporation of a random center effect to separate within- and between-center variance estimates. As participants will not be randomized to intervention arms, the proposed statistical analysis plan will also incorporate a multivariable modeling approach, with inclusion of potential confounders, to reduce bias in intervention effect estimates. Effect estimates will be reported with confidence intervals to convey variability in estimates.

Methods for sample size estimates were based on a simplified comparisons of means between the two arms (pre-post implementation periods). Necessary sample sizes were then inflated to account for multivariable model and to account for loss-to-follow-up, to ensure adequate power. The proposed sample size of 74 participants in the control period and 316 in the intervention period will provide at least 80-90% power to detect meaningful differences in mean Decisional Conflict Scale (DCS) score ranging from 5.0 to 7.7 units.

The impact of this study will be the creation of a model for integrating genetic testing into clinical practice that shows how to scale up genetic counseling services through the use of chatbots to deliver foundational information, and training nephrologists to deliver components of genetic counseling. Specifically, this model will demonstrate how to deliver APOL1 testing of live donor candidates, which can then be implemented across the country via implementation science approaches. The proposed study will prepare transplant programs to deliver culturally competent counseling coterminous with the completion of the NIH APOLLO study in ~5 years. The findings generated from this research have the potential to protect donor candidates' safety by improving their informed consent. As such, this proposal is timely and responsive to the NIDDK Program Announcement (PA-18-330) "Investigator-Initiated Clinical Trials Targeting Diseases within the Mission of NIDDK."

ELIGIBILITY:
Inclusion Criteria:

* Living kidney donor candidates who identify as African American/Black, Jamaican, Barbadian, Grenadian, Brazilian from Salvador Trinidadian, Panamanian, Honduran, Haitian, Garifunan, Palenque, Guyanese, Dominican, Peruvian, Belizean, and Native American, or state that they have African ancestry or are aware of having biologically-related family with African ancestry
* Living kidney donor candidates may be directed or non-directed donors
* Adults (ages 18+)
* English-speaking
* Cognitively intact individuals
* All genders

Exclusion Criteria:

* Individuals who do not identify as African American/Black and are not aware of having any biologically-related family with African ancestry and do not have African ancestry
* Only African Americans and people of African ancestry will be included because APOL1 risk variants are predominantly found in African Americans and people who have African ancestry.
* Pregnant women cannot be living kidney donors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | Day 1
  The Decisional Conflict Scale will measure donor candidates' perceived uncertainty in decision-making about donating and satisfaction with effective decision-making.
  Scores range from: 0-100 Higher scores reflect greater decisional conflict (a worse outcome).
Decisional Conflict Scale (DCS) | Approximately Day 7
  The Decisional Conflict Scale will measure donor candidates' perceived uncertainty in decision-making about donating and satisfaction with effective decision-making.
  Scores range from: 0-100 Higher scores reflect greater decisional conflict (a worse outcome).
Decisional Conflict Scale (DCS) | Approximately Day 30
  The Decisional Conflict Scale will measure donor candidates' perceived uncertainty in decision-making about donating and satisfaction with effective decision-making.
  Scores range from: 0-100 Higher scores reflect greater decisional conflict (a worse outcome).
Decisional Conflict Scale (DCS) | Approximately Day 60
  The Decisional Conflict Scale will measure donor candidates' perceived uncertainty in decision-making about donating and satisfaction with effective decision-making.
  Scores range from: 0-100 Higher scores reflect greater decisional conflict (a worse outcome).

SECONDARY OUTCOMES:
Preparation for Decision Making Scale (PDMS) Scores range from: Higher scores reflect greater preparation for decision making (a better outcome) | Day 1
  The Preparation for Decision Making Scale is a process measure that will assess donor candidates' perception of how useful the decision support intervention is in preparing them to communicate with their physician and make the donation about donating.
  Scores range from: 0-100 Higher scores indicate higher perceived level of preparation for decision making
Preparation for Decision Making Scale (PDMS) Scores range from: Higher scores reflect greater preparation for decision making (a better outcome) | Approximately Day 7
  The Preparation for Decision Making Scale is a process measure that will assess donor candidates' perception of how useful the decision support intervention is in preparing them to communicate with their physician and make the donation about donating.
  Scores range from: 0-100 Higher scores indicate higher perceived level of preparation for decision making
Preparation for Decision Making Scale (PDMS) Scores range from: Higher scores reflect greater preparation for decision making (a better outcome) | Approximately Day 30
  The Preparation for Decision Making Scale is a process measure that will assess donor candidates' perception of how useful the decision support intervention is in preparing them to communicate with their physician and make the donation about donating.
  Scores range from: 0-100 Higher scores indicate higher perceived level of preparation for decision making
Preparation for Decision Making Scale (PDMS) Scores range from: Higher scores reflect greater preparation for decision making (a better outcome) | Approximately Day 60
  The Preparation for Decision Making Scale is a process measure that will assess donor candidates' perception of how useful the decision support intervention is in preparing them to communicate with their physician and make the donation about donating.
  Scores range from: 0-100 Higher scores indicate higher perceived level of preparation for decision making
Willingness to Donate Scores range from: 0 to 10. Higher scores reflect greater willingness to donate. | Approximately Day 1
  This scale will assess how willing donor candidates are to donate.
  Scores range from 1-10 Higher scores reflect greater willingness to donate
Willingness to Donate Scores range from: 0 to 10. Higher scores reflect greater willingness to donate. | Approximately Day 7
  This scale will assess how willing donor candidates are to donate.
  Scores range from 1-10 Higher scores reflect greater willingness to donate
Willingness to Donate Scores range from: 0 to 10. Higher scores reflect greater willingness to donate. | Approximately Day 30
  This scale will assess how willing donor candidates are to donate.
  Scores range from 1-10 Higher scores reflect greater willingness to donate
Willingness to Donate Scores range from: 0 to 10. Higher scores reflect greater willingness to donate. | Approximately Day 60
  This scale will assess how willing donor candidates are to donate.
  Scores range from 1-10 Higher scores reflect greater willingness to donate
Satisfaction with the Informed Consent Process | Approximately Day 7
  This refers to donor candidates' decision-making quality, decision satisfaction, and perception of information.
  Scores range from: 1 - 5 Higher scores reflect greater satisfaction with the informed consent process
Satisfaction with the Informed Consent Process | Approximately Day 30
  This refers to donor candidates' decision-making quality, decision satisfaction, and perception of information.
  Scores range from: 1 - 5 Higher scores reflect greater satisfaction with the informed consent process
Satisfaction with the Informed Consent Process | Approximately Day 60
  This refers to donor candidates' decision-making quality, decision satisfaction, and perception of information.
  Scores range from: 1 - 5 Higher scores reflect greater satisfaction with the informed consent process

CONTACTS AND LOCATIONS:
Overall Officials: Elisa J Gordon, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JD, Agrawal A, Wicklund C, Duquette D, Friedewald J, Rasmussen LV, Gacki-Smith J, Tandon SD, Muhammad LN, Yancy CW, Dong S, Cooper M, Gilbert A, Shetty A, Gordon EJ. Implementation of a culturally competent APOL1 genetic testing programme into living donor evaluation: A two-site, non-randomised, pre-post trial design. BMJ Open. 2023 May 15;13(5):e067657. doi: 10.1136/bmjopen-2022-067657. PMID 37188469